CLINICAL TRIAL: NCT05507255
Title: Effect of Aerobic Exercise on Diurnal Cortisol Pattern in Premenstrual Syndrome: A Randomized Controlled Trial
Brief Title: Effect of Aerobic Exercise on Diurnal Cortisol Pattern in Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003807
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Premenstrual Syndrome
Keywords: Aerobic exercise; Relaxation training; Diurnal cortisol pattern; Premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation training (Active Comparator): Females will receive relaxation training, in the form of deep breathing, 3 days per week, for 8 weeks.
  Interventions: Other: Relaxation training
- The same relaxation training plus an aerobic exercise program (Experimental): Females will receive the same relaxation training, in addition to 30 minutes of a moderate aerobic exercise program on a treadmill, 3 days per week, for 8 weeks.
  Interventions: Other: Relaxation training; Other: An aerobic exercise program

INTERVENTIONS:
Other: Relaxation training — Relaxation training in the form of deep breathing exercises
Other: An aerobic exercise program — An aerobic exercise program of a moderate intensity, based on the target heart rate (THR) that will be calculated in accordance with Karvonen's equation, using resting heart rate (HRrest), maximal heart rate (HRmax) and training fraction. THR = HRrest (bpm) + (HRmax (bpm) - HRrest (bpm)) × training fraction.The exercise session will have three phases, warming up, active phase and cooling down.
  Arms: The same relaxation training plus an aerobic exercise program

SUMMARY:
The aim of this study will be to investigate the effect of aerobic exercise on diurnal cortisol pattern in premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual syndrome is manifested by recurrent emotional and depressive symptoms that may be associated with maladaptive coping with stress situations and the enhanced release of stress hormones, like cortisol hormone. Although previous studies revealed a flattened diurnal cortisol slope in women with PMS compared to healthy controls, there is no previous work on the effect of aerobic exercise on diurnal cortisol pattern in premenstrual syndrome. Therefore, this study will aim to investigate the effect of aerobic exercise participation on diurnal cortisol pattern in premenstrual syndrome.This trial will include two groups; group (A) will consist of 14 females who will receive relaxation training for 8 weeks, while group (B) will consist of 14 females who will receive the same relaxation training along with aerobic exercise for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary, virginal, adult, non-smoker females suffering from premenstrual syndrome.
2. They should have regular menstrual cycles (cycles of 21-35 days with a bleeding time of 3-10 days)
3. They should have the following criteria in daily record of severity of problems in at least one of two consecutive menstrual cycles prior to treatment starting to confirm premenstrual syndrome diagnosis: a) more than three items have an average score over 3 during the luteal phase, and b) a luteal phase score is 30% more than a follicular phase score.
4. No traumatic life events in the last 2 months before starting the study.
5. Their age will be 18-23 years
6. Their body mass index (BMI) will be less than 30 kg/m2.

Exclusion Criteria:

1. Menstrual problems (e.g. menorrhagia, metrorhagia and polycystic ovary disease).
2. Cardio-respiratory, renal, neurological and pelvic inflammatory diseases, tumors, infections, anemia, diabetes, hypertension, asthma, rheumatoid arthritis, headache, migraine, thyroid or mental disorders.
3. Participation at any other exercise training program during this study.
4. Receiving any kind of medications, hormonal treatment or supplementation (vitamin, mineral or herbal supplement).

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Diurnal cortisol pattern | 8 weeks
  It will be evaluated through calculating the ratio of morning cortisol level to evening cortisol level for all participants at baseline and after 8 weeks of treatment.
Severity of premenstrual symptoms | 8 weeks
  Severity of premenstrual symptoms of all participants will be measured through daily record of severity of problems (DRSP) at baseline and after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Osman, Principal Investigator — Department of Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt